CLINICAL TRIAL: NCT04093583
Title: Randomized Clinical Trial, Conventional Treatment-controlled, Studying the Efficacy of Plasma Rich in Growth Factor (PRGF®) in Alveolar Ridge Preservation After Simple Exodontia in the Anterior Region of Maxilla.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIBEA_04_EC_19_ALV; 2019-001167-75 (EudraCT Number)
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dental Implantation
Keywords: exodontia; PRGF; alveolar ridge preservation
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simple suture (Active Comparator)
  Interventions: Procedure: Exodontia
- PRGF-Endoret (Experimental)
  Interventions: Procedure: Exodontia; Drug: Alveolar ridge preservation with a PRP (PRGF-Endoret); Device: Preparation of PRGF using Endoret technology

INTERVENTIONS:
Procedure: Exodontia — Atraumatic exodontia followed by simple suture
Drug: Alveolar ridge preservation with a PRP (PRGF-Endoret) — Filling of the alveolus with PRGF clot and fibrin plug.
  Arms: PRGF-Endoret
Device: Preparation of PRGF using Endoret technology — Preparation of PRGF using Endoret technology following manufacturer instructions
  Arms: PRGF-Endoret

SUMMARY:
This RCT aims to study the efficacy and safety of PRGF-Endoret in alveolar ridge preservation in the aesthetic zone. The control group is the spontaneous healing occuring after the suturing of the alveolus. The primary endpoint is the bone regeneration measured in biopsies obtained from the regenerated alveolar bone.

ELIGIBILITY:
Inclusion Criteria:

* - Subjects of both sexes with an age greater than or equal to 18 years.
* Clinical indication for a simple exodontia in the aesthetic zone (from left 2nd premolar to the right 2nd premolar in the maxilla).
* Need of a dental implant placement in the extraction site.
* Availability to follow-up during the treatment period
* Subjects with non-active periodontal disease.
* Buccal dehiscence < than 25% in the vestibular table

Exclusion Criteria:

* - Presence of an active infection
* Loss of any plate of the socket
* Severe inflammation in the area of the exodontia previous to the intervention
* Have previous diagnosis of a coagulopathy.
* Have previous diagnosis of any autoinmune disease.
* Have received radiotherapy, chemotherapy or immunosuppressive treatments, systemic corticosteroids and/or anticoagulants the 30 days prior to inclusion
* Regular treatment with AINES or other antiinflammatory drugs
* Previous history of chronic hepatitis or heatic cirrhosis
* Positive markers for VHC, AgHBs, VIH I/II or Treponema pallidum
* Uncontrolled diabetes mellitus (Glycosylated hemoglobin higher than 9%)
* Subjects submitted to hemodyalisis
* Presence of malignant tumour, haemangiomas or angioma in the exodontia region.
* Previous history of ischemic cardiopathy in the last year.
* Pregnancy or womens in childbearing age who do not take contraception measures.
* Nursing womens
* Metabolic bone disease
* Ongoing treatment with biphosphonates both through oral or intravenous administration
* Smoking habits (> 10 cigarrettes/day)
* In general, any disability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Bone regeneration | 12 months
  Quantity of new bone measured in bone biopsies obtained after alveolar ridge preservation

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Eduardo Anitua Private Clinic, Vitoria-Gasteiz, Alava
  - Clinica dental Murias, Getxo, Bizkaia
  - Clinica Dental Loroño, Galdakao, Viscay
  - Clinica Ereaga, Getxo, Viscay
  - Clínica Dental González Mosquera, A Coruña